CLINICAL TRIAL: NCT04276571
Title: EMPATIA@Lecco- Balance Rehabilitation of Autistic Children With Virtual rEality
Acronym: BRAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIP-679
Record Dates: First submitted 2020-02-18; First posted 2020-02-19 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Autism Spectrum Disorder
Keywords: motor abilities
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GRAIL (Experimental)
  Interventions: Device: exergames with GRAIL virtual immersive reality environment
- No treatment (No Intervention)

INTERVENTIONS:
Device: exergames with GRAIL virtual immersive reality environment — The participants will perform exergames on GRAIL immersive virtual reality to improve balance (e.g. load shifts, exercises with adaptations to motor perturbations). GRAIL can provide proprioceptive and visual feedback to participants.
  Arms: GRAIL

SUMMARY:
The general objective of this project is to investigate the possible efficacy of a training based on proprioceptive and visual feedback carried out with the GRAIL (Motekforce Link) virtual reality environment on postural control and balance skills of school-aged children with clinical diagnosis of ASD.

ELIGIBILITY:
Inclusion Criteria:

* a clinical diagnosis of ASD
* All participants were required to have estimated FSIQ of 80 or above

Exclusion Criteria:

* using any stimulant or non-stimulant medication that affects the central nervous system
* having an identified genetic disorder
* having vision or hearing problems
* suffering from chronic or acute medical illness
* presence of epilepsy

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
experimental balance assessment | approximately 6 weeks after starting the intervention
  Balance assessment through the evaluation (with both open and closed eyes) of the center of pression using the GRAIL platform
Movement Assessment Battery for Children 2 (MABC2) (Henderson et al., 2007). | approximately 6 weeks after starting the intervention
  The MABC2 consists of eight subtests that evaluate three components of motor proficiency: manual dexterity, ball skills, and static and dynamic balance. For the MABC2, higher scores are indicative of better motor performance.

SECONDARY OUTCOMES:
Developmental Coordination Disorder Questionnaire (DCDQ) (Wilson et al., 2007). | approximately 6 weeks after starting the intervention
  The DCDQ is a 15-item questionnaire that investigates gross and fine motor skill impairments. The DCDQ yields a raw total score (score range 15-75); higher scores indicate better motor functioning as rated by the parents.
assessment of balance in response to perturbation applied by accelerating the dual-belt treadmill the dominant side at toe-off | approximately 6 weeks after starting the intervention
  assessment of balance in response to perturbation applied by accelerating the dual-belt treadmill
assessment of overground balance using GSENSOR (BTS Bioengineering), a medical device for motion analysis | approximately 6 weeks after starting the intervention
  assessment of overground balance using GSENSOR (BTS Bioengineering), a medical device for motion analysis
evaluation of gait features using the GRAIL (Motekforce Link) | approximately 6 weeks after starting the intervention
  evaluation of gait features using the GRAIL (Motekforce Link)

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Institute IRCCS E. Medea, Bosisio Parini, Lecco, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Biffi E, Costantini C, Ceccarelli SB, Cesareo A, Marzocchi GM, Nobile M, Molteni M, Crippa A. Gait Pattern and Motor Performance During Discrete Gait Perturbation in Children With Autism Spectrum Disorders. Front Psychol. 2018 Dec 11;9:2530. doi: 10.3389/fpsyg.2018.02530. eCollection 2018. PMID 30618953
- [Derived] Falivene A, Scaccabarozzi G, Busti Ceccarelli S, Molteni M, Klingels K, Verbecque E, Storm FA, Biffi E, Crippa A. Virtual Reality-Based Postural Balance Training in Autistic Children: A Pilot Randomized Controlled Trial. J Clin Med. 2025 Aug 8;14(16):5616. doi: 10.3390/jcm14165616. PMID 40869441